CLINICAL TRIAL: NCT03667053
Title: Phase 3, Randomized, Double-blind, Placebo/Active-controlled, Parallel-arm Trial to Assess Efficacy, Safety, and Pharmacokinetics of Dasiglucagon Relative to Placebo/GlucaGen® as Rescue Therapy for Severe Hypoglycemia in Children With T1DM Treated With Insulin
Brief Title: Trial to Confirm the Efficacy and Safety of Dasiglucagon in the Treatment of Hypoglycemia in T1DM Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP4207-17086
Record Dates: First submitted 2018-09-07; First posted 2018-09-12 (Actual); Results first posted 2021-05-10 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-05

CONDITIONS: Hypoglycemia
Keywords: Glucagon; Dasiglucagon
MeSH Terms: conditions — Hypoglycemia | interventions — dasiglucagon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- dasiglucagon (Experimental): Single fixed dose (s.c.injection) of dasiglucagon
  Interventions: Drug: dasiglucagon
- placebo (Placebo Comparator): Single fixed dose (s.c.injection) of placebo
  Interventions: Drug: placebo
- GlucaGen® (Active Comparator): Single fixed dose (s.c.injection) of GlucaGen®
  Interventions: Drug: GlucaGen HypoKit

INTERVENTIONS:
Drug: dasiglucagon — glucagon analog
  Other Names: ZP4207
  Arms: dasiglucagon
Drug: placebo — placebo for dasiglucagon
  Other Names: placebo for dasiglucagon
  Arms: placebo
Drug: GlucaGen HypoKit — native glucagon
  Arms: GlucaGen®

SUMMARY:
A phase 3, randomized, double-blind, placebo- and active-controlled, parallel-arm trial to assess the efficacy, safety, and pharmacokinetics of dasiglucagon relative to placebo and GlucaGen® when administered as a rescue therapy for severe hypoglycemia in children with type 1 diabetes mellitus (T1DM) treated with insulin

DETAILED DESCRIPTION:
At least 40 children ≥6 years and <18 years of age with T1DM were planned to be randomized into the trial (2:1:1 for dasiglucagon:placebo:GlucaGen) and stratified by age intervals: 6 years to <12 years, and 12 years to <18 years; and by injection site (abdomen or thigh). A minimum of 16 patients were enrolled into each age group, including a minimum of 8 patients in each age group in the dasiglucagon treatment arm. In Germany only, a staggered approach was applied, whereby a positive safety assessment needed to be available for at least 10 patients in the age group of 12 years to <18 years who had completed the dosing visit in the overall trial before younger patients (6 to 11 years of age) were allowed to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Following receipt of verbal and written information about the trial, patient, parent(s) or guardian(s) of the patient must provide signed informed consent before any trial-related activity is carried out
2. Female or male patients with T1DM for at least 1 year, diagnostic criteria as defined by the American Diabetes Association; and receiving daily insulin
3. At least 6.0 years of age (inclusive) and less than 18.0 years
4. Body weight ≥20 kg
5. Female patients must meet one of the following criteria:

   a. Participant is of childbearing potential and agrees to use one of the accepted contraceptive regimens throughout the entire duration of the trial from screening until last follow-up visit. An acceptable method of contraception includes at least one of the following: i. Abstinence from heterosexual intercourse ii. Systemic contraceptives (birth control pills, injectable/implant/ insertable hormonal birth control products, transdermal patch); if the participant is using systemic contraceptives, she must use an additional form of acceptable contraception (iii or iv, below) iii. Intrauterine device (with and without hormones) iv. Condom with spermicide or b. Participant is of non-childbearing potential due to pre-puberty status or a medical condition confirmed by the investigator
6. Male patients must meet the following criteria: If sexually active, uses condom and partner practices contraception during the trial from screening and until last follow-up visit
7. Willingness to adhere to the protocol requirements

   -

   Exclusion Criteria:

1. Females who are pregnant according to a positive urine pregnancy test, actively attempting to get pregnant, or are lactating 2. Known or suspected allergy to trial product(s) or related products 3. History of anaphylaxis or symptoms of severe systemic allergy (such as angioedema) 4. Previous randomization in this trial 5. History of an episode of severe hypoglycemia that required a third party assistance within a month prior to screening visit 6. History of hypoglycemic events associated with seizures or hypoglycemia unawareness in the last year prior to screening 7. History of epilepsy or seizure disorder 8. Receipt of any investigational drug within 3 months prior to screening 9. Active malignancy within the last 5 years 10. Congestive heart failure, New York Heart Association class II-IV 11. Current bleeding disorder, including anti-coagulant treatment 12. Known presence or history of pheochromocytoma (i.e. adrenal gland tumor) or insulinoma (i.e. insulin secreting pancreas tumor) 13. Use of a daily systemic beta-blocker drug, indomethacin, warfarin or anticholinergic drugs in the previous 28 days before Day 1 of this trial 14. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 × the upper limit of the normal range (ULN), bilirubin >1.5 × ULN, estimated glomerular filtration rate <30 mL/min/1.73 m2 according to the Modification of Diet in Renal Disease study definition, or altered electrolyte values of clinical relevance for cardiac conduction, as judged by the investigator 15. Clinically significant abnormal electrocardiogram (ECG) at screening as judged by the investigator 16. Clinically significant illness within 4 weeks before screening, as judged by the investigator 17. Surgery or trauma with significant blood loss within the last 2 months prior to screening 18. Patients with mental incapacity or language barriers which preclude adequate understanding or cooperation, who are unwilling to participate in the trial, or who in the opinion of the investigator should not participate in the trial 19. Any condition interfering with trial participation or evaluation or that could be hazardous to the patient 20. The use of prescription or non-prescription medications known to cause QT prolongation

-

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Sylvest, MSc Pharm, Study Director — Zealand Pharma A/S
Locations (5):
- United States (3):
  - AMCR Institute, Inc, Escondido, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Indiana University, Department of Pediatrics, Indianapolis, Indiana
- Auf der Bult - Diabetes Center for Children, Hanover, Germany
- University Medical Center Ljubljana, Children's Hospital, Department for Endocrinology, Diabetes and Metabolism, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasiglucagon 0.6 mg: Single fixed dose (subcutaneous injection) of dasiglucagon
  dasiglucagon: glucagon analog
- Placebo: Single fixed dose (subcutaneous injection) of placebo
  placebo: placebo for dasiglucagon
- GlucaGen® 1.0 mg: Single fixed dose (subcutaneous injection) of GlucaGen® (0.5 mg if body weight <25 kg)
  GlucaGen HypoKit: native glucagon
Period: Overall Study
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Started (Randomized subjects) | 21 | 11 | 10
Randomized and Treated | 20 | 11 | 10
Completed | 20 | 11 | 10
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set of all randomized and treated participants. Treatment assignment was based on the treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg | Total
Number analyzed (Participants) | 20 | 11 | 10 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 11 | 10 | 41
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.3 (3.42) | 12.8 (3.25) | 12.4 (3.50) | 12.5 (3.32)
Age, Customized [Count of Participants; unit: Participants]
  Age 6-11 years | 8 | 4 | 4 | 16
  Age 12-17 years | 12 | 7 | 6 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 2 | 18
  Male | 10 | 5 | 8 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 1 | 7
  Not Hispanic or Latino | 16 | 8 | 9 | 33
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 19 | 10 | 10 | 39
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 9 | 7 | 29
  Slovenia | 6 | 2 | 3 | 11
  Germany | 1 | 0 | 0 | 1
Body weight [Mean (Standard Deviation); unit: kg] | 51.54 (22.202) | 54.95 (21.404) | 48.81 (14.992) | 51.79 (20.106)
Body mass index [Mean (Standard Deviation); unit: kg per square meter] | 20.74 (6.057) | 20.39 (4.885) | 18.92 (2.617) | 20.20 (5.050)

OUTCOME MEASURES:

1. Primary Outcome: Time to Plasma Glucose Recovery
Description: Plasma glucose recovery was defined as first increase in plasma glucose of ≥20 mg/dL (1.1 mmol/L) from baseline during the hypoglycemic clamp procedure without administration of rescue intravenous (IV) glucose. Patients who received rescue IV glucose before 45 minutes and patients not recovering within 45 minutes after dosing were censored at 45 minutes. Time to plasma glucose recovery was summarized for each treatment group using Kaplan Meier (KM) estimates together with the 95% confidence interval.
  Note that the upper confidence limit for the placebo median was not estimable, but is set to 45 minutes (censored value) here.
Time Frame: 0-45 minutes after dosing
Population: Full analysis set (same as the safety analysis set) of all randomized and treated patients. Treatment assignment was based on the randomized treatment. Assignment to the stratification factor injection site was based on the planned and not the actual used injection site.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 11 | 10
minutes | 10.00 [8.00 to 12.00] | 30.00 [20.00 to 45.00] | 10.00 [8.00 to 12.00]
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs Placebo; The treatment group difference between dasiglucagon and placebo was evaluated inferentially using a pairwise two-sided log rank test stratified by injection site and age group; Test type: Superiority; p < 0.001, Log Rank

2. Secondary Outcome: Plasma Glucose Recovery
Description: Plasma glucose recovery within 30 minutes, within 20 minutes, within 15 minutes, and within 10 minutes after study drug injection without administration of rescue intravenous (IV) glucose. Plasma glucose recovery was defined as the first increase in plasma glucose of ≥20 mg/dL (1.1 mmol/L) from baseline without administration of rescue intravenous glucose.
Time Frame: 0-30 minutes after dosing: assessed at 10, 15, 20 and 30 minutes after study drug injection
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 11 | 10
Participants
  Glucose recovery at 30 minutes | 20 | 6 | 10
  Glucose recovery at 20 minutes | 20 | 2 | 10
  Glucose recovery at 15 minutes | 19 | 0 | 10
  Glucose recovery at 10 minutes | 13 | 0 | 6
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs Placebo; The recovery rates of dasiglucagon and placebo were compared at each time point using a Cochran-Mantel-Haenszel test stratified by age group and injection site. Testing followed an a priori defined hierarchical inferential test order, proceeding until the first failure to reject the null hypothesis comparing dasiglucagon versus placebo; Test type: Superiority; p = 0.0073, Cochran-Mantel-Haenszel — Assessed at 30 minutes. Note that p-value was 0.0005 at 10 minutes and <0.0001 at 15 and 20 minutes

3. Secondary Outcome: Plasma Glucose Changes From Baseline
Description: Plasma glucose changes from baseline within 30 minutes, within 20 minutes, within 15 minutes, and within 10 minutes after trial product injection or at the time of rescue intravenous (IV) glucose
Time Frame: 0-30 minutes after dosing: assessed at 10, 15, 20 and 30 minutes after study drug injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 11 | 10
mg/dL
  At 30 minutes | 98.459 (19.6527) | 17.510 (15.6313) | 85.225 (12.5052)
  At 20 minutes | 65.369 (15.2461) | 7.322 (13.3543) | 58.000 (10.5297)
  At 15 minutes | 45.342 (15.0860) | 0.835 (11.1276) | 40.631 (9.7317)
  At 10 minutes | 27.225 (13.6768) | -3.405 (8.0276) | 20.919 (6.7227)
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs Placebo; Change from baseline in plasma glucose at 30, 20, 15, and 10 minutes after investigational product injection was calculated using nominal sampling times and analyzed using an analysis of variance model with treatment, age group and injection site for each endpoint. Testing followed an a priori defined hierarchical inferential test order, proceeding until the first failure to reject the null hypothesis comparing dasiglucagon versus placebo; Test type: Superiority; p < 0.0001, ANOVA — The p-value was <0.0001 at all time points (10, 15, 20 and 30 minutes)

4. Secondary Outcome: Pharmacodynamics - Area Under the Effect Curve (0-30 Minutes)
Description: Plasma glucose response as area under the effect curve above baseline from time 0 to 30 minutes (AUE0-30min). Plasma glucose was determined at pre-dose and at 4, 6, 8, 10, 12, 15, 17, 20, 30, and 45 minutes (and at 60 minutes if the patient weighed ≥21 kg) after dosing.
Time Frame: 0-30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol*h/L
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 11 | 10
mmol*h/L | 22.83 (6.126) | 1.81 (4.641) | 19.66 (3.410)

5. Secondary Outcome: Administration of Rescue IV Glucose Infusion After IMP Injection
Description: Number of patients receiving IV rescue glucose administration for hypoglycemia after administration of IMP. IV = intravenous. IMP = investigational medicinal product.
Time Frame: 0-45 minutes
Population: Safety analysis set (same as the full analysis set) of all randomized and treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 11 | 10
Participants | 0 | 1 | 0

6. Secondary Outcome: Time to First IV Glucose Infusion After IMP Administration
Description: Time to first IV rescue glucose administration for hypoglycemia after administration of IMP. IV = intravenous. IMP = investigational medicinal product.
Time Frame: 0-45 minutes
Population: Only the patient who received IV glucose administration is included.
Measure: Number; unit: minutes
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Number analyzed (Participants) | 0 | 1 | 0
minutes |  | 12 |

7. Secondary Outcome: Pharmacokinetics: AUC0-30 Min
Description: Area under the plasma dasiglucagon or GlucaGen concentration versus time curve from 0 to 30 minutes post-dose. Samples were collected before dosing and at 10, 20, 30, 40, 60, 90, 140, 220, and 300 minutes after dosing.
Time Frame: 0-30 minutes
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pmol/L
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 10
h*pmol/L | 376 (78.1) | 376 (63.3)

8. Secondary Outcome: Pharmacokinetics: AUC0-300min
Description: Area under the plasma dasiglucagon or GlucaGen concentration versus time curve from 0 to 300 minutes post-dose. Samples were collected before dosing and at 10, 20, 30, 40, 60, 90, 140, 220, and 300 minutes after dosing.
Time Frame: 0-300 minutes
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pmol/L
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 10
h*pmol/L | 1810 (44.8) | 1370 (72.7)

9. Secondary Outcome: Pharmacokinetics: AUC0-inf
Description: Area under the plasma dasiglucagon or GlucaGen concentration versus time curve from 0 to infinitely post-dose. Samples were collected before dosing and at 10, 20, 30, 40, 60, 90, 140, 220, and 300 minutes after dosing.
Time Frame: 0-300 minutes
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pmol/L
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 10
h*pmol/L | 1850 (45.1) | 1530 (70.3)

10. Secondary Outcome: Pharmacokinetics: Cmax
Description: Maximum of all valid plasma dasiglucagon or GlucaGen concentration measurements from 0 to 300 minutes post-dose. Samples were collected before dosing and at 10, 20, 30, 40, 60, 90, 140, 220, and 300 minutes after dosing.
Time Frame: 0-300 minutes
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 10
pmol/L | 1160 (61.2) | 1120 (80)

11. Secondary Outcome: Pharmacokinetics: Tmax
Description: Time to maximum of plasma dasiglucagon or GlucaGen concentration measurements. Samples were collected before dosing and at 10, 20, 30, 40, 60, 90, 140, 220, and 300 minutes after dosing.
Time Frame: 0-300 minutes
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 10
hours | 0.35 [0.167 to 1.5] | 0.333 [0.167 to 0.5]

12. Secondary Outcome: Pharmacokinetics: λz
Description: Terminal elimination rate constant of plasma dasiglucagon or GlucaGen. Samples were collected before dosing and at 10, 20, 30, 40, 60, 90, 140, 220, and 300 minutes after dosing.
Time Frame: 0-300 minutes
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 10
1/hour | 1.11 (37.4) | 0.504 (27.2)

13. Secondary Outcome: Pharmacokinetics: t½
Description: Terminal plasma elimination half-life of dasiglucagon or GlucaGen. Samples were collected before dosing and at 10, 20, 30, 40, 60, 90, 140, 220, and 300 minutes after dosing.
Time Frame: 0-300 minutes
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 10
hours | 0.623 (37.4) | 1.38 (27.2)

14. Secondary Outcome: Pharmacokinetics: CL/f
Description: Total body clearance of plasma dasiglucagon or GlucaGen. Samples were collected before dosing and at 10, 20, 30, 40, 60, 90, 140, 220, and 300 minutes after dosing.
Time Frame: 0-300 minutes
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 10
L/h | 96.1 (45.1) | 188 (70.3)

15. Secondary Outcome: Pharmacokinetics: Vz/f
Description: Volume of distribution of plasma dasiglucagon or GlucaGen. Samples were collected before dosing and at 10, 20, 30, 40, 60, 90, 140, 220, and 300 minutes after dosing.
Time Frame: 0-300 minutes
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: litres
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 10
litres | 86.4 (62.2) | 373 (81.1)

16. Secondary Outcome: Pharmacokinetics: MRT
Description: Mean residence time of plasma dasiglucagon or GlucaGen. Samples were collected before dosing and at 10, 20, 30, 40, 60, 90, 140, 220, and 300 minutes after dosing.
Time Frame: 0-300 minutes
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 20 | 10
hours | 1.27 (29.5) | 1.86 (21.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first trial-related activity after the patient had signed the informed consent to the end of the follow-up period (28 days).
Groups:
- Age Group 6-11 Years - Dasiglucagon: Patients in the dasiglucagon group in the age group 6-11 years
- Age Group 6-11 Years - Placebo: Patients in the placebo group in the age group 6-11 years
- Age Group 6-11 Years - GlucaGen: Patients in the GlucaGen group in the age group 6-11 years
- Age Group 12-17 Years - Dasiglucagon: Patients in the dasiglucagon group in the age group 12-17 years
- Age Group 12-17 Years - Placebo: Patients in the placebo group in the age group 12-17 years
- Age Group 12-17 Years - Glucagen: Patients in the GlucaGen group in the age group 12-17 years
- Dasiglucagon 0.6 mg: Full population. Single fixed dose (subcutaneous injection) of dasiglucagon
- Placebo: Full population. Single fixed dose (subcutaneous injection) of placebo
- GlucaGen® 1.0 mg: Full population. Single fixed dose (subcutaneous injection) of GlucaGen® (0.5 mg if body weight <25 kg)
Arm/Group | Age Group 6-11 Years - Dasiglucagon | Age Group 6-11 Years - Placebo | Age Group 6-11 Years - GlucaGen | Age Group 12-17 Years - Dasiglucagon | Age Group 12-17 Years - Placebo | Age Group 12-17 Years - Glucagen | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4 | 0/4 | 0/12 | 0/7 | 0/6 | 0/20 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4 | 0/4 | 0/12 | 0/7 | 0/6 | 0/20 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 3/8 | 1/4 | 4/4 | 12/12 | 6/7 | 5/6 | 15/20 | 7/11 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Group 6-11 Years - Dasiglucagon (N=8) | Age Group 6-11 Years - Placebo (N=4) | Age Group 6-11 Years - GlucaGen (N=4) | Age Group 12-17 Years - Dasiglucagon (N=12) | Age Group 12-17 Years - Placebo (N=7) | Age Group 12-17 Years - Glucagen (N=6) | Dasiglucagon 0.6 mg (N=20) | Placebo (N=11) | GlucaGen® 1.0 mg (N=10)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Injection site edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 11 (12) | 0 (0) | 1 (1) | 13 (14) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 8 (11) | 0 (0) | 0 (0) | 10 (13) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (16) | 2 (2) | 2 (2) | 4 (16) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT03667053/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT03667053/SAP_001.pdf